CLINICAL TRIAL: NCT05863637
Title: Anxiety Treatment in Primary Care: an Evaluation of Intensive Dynamic Short-term Therapy
Brief Title: Intensive Short-Term Dynamic Psychotherapy (ISTDP) for Anxiety Diagnoses in a Primary Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Linnaeus University (Other)
Collaborators: Kalmar County Hospital (Other)
Responsible Party: Principal Investigator, Suzanne Petersson, PhD, Linnaeus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LinnaeusUSP
Record Dates: First submitted 2023-04-27; First posted 2023-05-18 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Psychotherapy; Anxiety Disorders; Psychiatric &or Mood Disorder
Keywords: Anxiety Disorders; Primary Care Setting; Psychotherapy; Clinical Research
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Controlled study; participants (e.g. primary care patients with an anxiety disorder) will be recruited consecutively to the study, they will be put on a waiting-list for 3 months (= standard procedure) and thus be their own control person.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated (Experimental): Participants are their own controls when they are on the waiting list before treatment, and they will later be treated with the ISTDP.
  Interventions: Other: Intensive Short-Term Dynamic Psychotherapy

INTERVENTIONS:
Other: Intensive Short-Term Dynamic Psychotherapy — A dynamic and intensive psychotherapy with eight therapeutic sessions

SUMMARY:
Living with anxiety often means great suffering for the person affected. The trend points to a continued increase in anxiety problems in the population, especially in the 18-44 age group. Inadequate treatment of this condition can lead to long-term sick leave, isolation, exclusion and, in the worst case, to death. The treatment methods that are available in primary care today help some but far from all. Therefore, the investigators want to scientifically evaluate a shorter version of a proven emotion-focused psychotherapy in order to increase the treatment range for this patient group. The aim of this project is to, in a primary care setting, test and evaluate an intensive, emotion-focused short-term therapy, ISTDP (Intensive Short-Term Dynamic Psychotherapy) for patients with an anxiety diagnosis. The method is well-proven on patients with more severe mental conditions (personality disorders) with good results, but the treatment has only been tested to a limited extent on patients with anxiety symptoms. The investigators want to investigate the effectiveness of treating various anxiety states for primary care patients. The treatment is expected to provide an addition to today's methods, which overall will provide better treatment results for this, increasing in number, group of patients who often seek primary care.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care patients with primary anxiety diagnoses at a Health Care clinic in Sweden. Sufficient language competence in Swedish is required of the participants to understand, read, speak and write.

Exclusion Criteria:

* Major reading-writing and learning difficulties, severe psychiatric problems such as psychosis, eating disorder, current major depression, recurrent depression, severe trauma, acute crisis reaction, exhaustion, acute risk of suicide (assessed according to the suicide scale), addiction.
* Diagnosed specific phobia or obsessive-compulsive disorder that must be primarily treated with CBT. Concurrent psychological treatment, anxiety-relieving medication such as benzodiazepines, or recently started antidepressant treatment (< 3 months of treatment) are also exclusion criteria for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Generalized Anxiety Disorder-7 (GAD-7) scorings | Changes in scorings from baseline scorings to scorings after 9-10 months.
  Self-report measure. The GAD-7 consists of 7 items which are scored 0-3, with a total score ranging from 0-21. Higher scores correspond to worse outcome.
  measures

SECONDARY OUTCOMES:
The Perceived Health Questionnaire (PHQ-9) scorings | Changes in scorings from baseline scorings to scorings after 9-10 months.
  Self-report measure. The PHQ-9 consists of 9 items, which are scored from 0-3 and a total score ranging from 0-27. Higher scores correspond to worse outcome.
The Panic Disorder Severity Scale (PDSS) scorings | Changes in scorings from baseline scorings to scorings after 9-10 months.
  Self-report measure. The PDSS consists of 7 items, which are scored from 0-4, with a total score ranging from 0-28. Higher scores correspond to worse outcome.
The Brunnsvikens Brief Quality of Life Inventory (BBQ) scorings | Changes in scorings from baseline scorings to scorings after 9-10 months.
  Self-report measure. The BBQ has a total of 12 items covering 6 life areas. Possible total score range is 0-96. Higher scores correspond to a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Fagerström, Professor, Study Director — Director of the Research Board in Region Kalmar
Locations (1):
- Region Kalmar, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No